CLINICAL TRIAL: NCT03459209
Title: Effect of Different Tube-feeding Techniques on the Delivery of Human Milk Long-chain Polyunsaturated Fatty Acids
Brief Title: Effect of Tube Feeding on LCPUFAs Delivery
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, Associate Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: SO-2017-LCPUFA
Record Dates: First submitted 2018-03-03; First posted 2018-03-08 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Lipid Depletion; Human Milk; Tube Feeding
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human milk samples (17 specimens)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: tube feeding — The obtained milk aliquots undergo in vitro administration through three different tube feeding techniques.

SUMMARY:
Long-chain polyunsaturated fatty acids (LCPUFAs) docosahexaenoic (DHA) arachidonic acid (AA) are major building blocks for the lipid bilayer of neuronal and retinal membranes and play a crucial role in brain and visual development. Humans lack enzymes synthetizing DHA and AA precursors and thus rely upon dietary sources to achieve adequate intakes. Human milk (HM) feeding, either own mother's milk (OMM) or donor milk (DM), is the first nutritional choice for preterm infants and provides appropriate LCPUFAs amounts to support neurological and visual development of this fragile population.

Due to their immaturity, preterm infants are often unable to coordinate sucking and swallowing, thus requiring tube feeding (TF) for prolonged time periods. During TF, fatty acids tend to separate from aqueous milk components and to adhere to the infusion set, thus reducing the delivery of HM lipid contents. To dare, however, a targeted evaluation of TF-related LCPUFAs losses has not been performed.

This study aims to quantitatively assess, by means of gas chromatography coupled to mass spectrometry, the effect of bolus and different continuous feeding methods routinely adopted for preterm infants' enteral nutrition on the delivery of DHA and AA contained in human milk samples.

DETAILED DESCRIPTION:
Despite recent improvements in neonatal care, the delicate extra-uterine maturation of central nervous system place preterm infants at high risk for neurodevelopmental impairment.

Long-chain polyunsaturated fatty acids (LCPUFAs) docosahexaenoic (DHA, 22:6 n-3) and arachidonic acid (AA, 20:4 n-6) are major building blocks for the lipid bilayer of neuronal and retinal membranes, thus playing a crucial role in brain and visual development. Humans, however, lack enzymes for synthetizing n-3 and n-6 precursors of DHA and AA, thus strictly relying upon dietary sources. Human milk (HM) feeding, either own mother's milk (OMM) or donor milk (DM), is the first nutritional choice for preterm infants and, if maternal dietary intakes are adequate, is expected to provide appropriate LCPUFAs amounts in this fragile population. Nevertheless, in addition to the type of milk, equal attention should be paid to its delivery methods.

Due to their immaturity, preterm infants are often unable to coordinate sucking and swallowing, thus requiring tube feeding (TF) for prolonged time periods. During TF, fatty acids tend to separate from aqueous milk components and to adhere to the infusion set, thus reducing the delivery of HM lipid contents. To dare, however, a targeted evaluation of TF-related LCPUFAs losses has not been performed.

This study aims to quantitatively assess the effect of different TF techniques routinely adopted for preterm infants' enteral nutrition on DHA and AA delivery.

Mothers of preterm infants (≤32 weeks' gestation) admitted to the Neonatal Intensive Care Unity of Sant'Orsola-Malpighi University Hospital, Bologna (Italy), and HM donors adhering to the Human Milk Bank of Bologna will be enrolled in the present study if written, informed consent to participate will be obtained.

Samples of fresh human milk or pasteurized donor milk, each one of 65 ml, will be collected. These samples will be then split into three 20-ml aliquots that will be subjected to as many TF modalities, whereas the remaining 5 ml will serve as baseline.

By using a 20-ml polypropylene syringe connected to a feeding tube, three different TF modalities will be simulated at room temperature conditions: gravity bolus feeding (BF), horizontal continuous feeding (HCF) and 45-degree-angled continuous feeding (ACF).

HCF and ACF will be delivered over 3 hours. During HCF the feeding syringe will be horizontal, whereas during ACF the tip of the feeding syringe will be angled 45° upward from the longitudinal axis. Moreover, in order to evaluate the efficacy of lipid delivery in relation to different phases of continuous feeding, HM delivered from 0 to 90 min and from 91 to 180 min will be collected and analyzed separately.

Eventually, LCPUFAs contents in the resulting specimens will be analyzed by means of gas chromatography coupled to mass spectrometry (GC-MS) at the laboratory of the Center for Applied Biomedical Research (CRBA) of S. Orsola-Malpighi University Hospital in Bologna, Italy.

ELIGIBILITY:
Inclusion Criteria:

* Availability of breast milk
* Stage of lactation: between 2 to 3 months after delivery
* Written, informed consent obtained

Exclusion Criteria:

* breast milk not available
* <2 months or >3 months from delivery
* no consent obtained

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breastfeeding mothers of preterm infants (≤32 weeks gestation) admitted to the Neonatal Intensive Care Unity of Sant'Orsola-Malpighi University Hospital, Bologna (Italy) and human milk donors adhering to the Human Milk Bank of Bologna.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
LCPUFA loss | 3 hours
  Reduction in DHA and/or AA contents of each human milk aliquot after tube feeding administration

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Corvaglia, MD, Principal Investigator — Sant'Orsola-Malpighi University Hospital, Bologna
Locations (1):
- Neonatal Intensive Care Unit, S.Orsola-Malpighi Hospital, Bologna, Italy